CLINICAL TRIAL: NCT01684358
Title: A Randomized Controlled Trial on the Effect of Sino-implant (II) Use on Condom Use Among Women in Kingston, Jamaica
Brief Title: A Trial on the Effect of Sino-implant (II) Use on Condom Use Among Women in Kingston, Jamaica
Acronym: SIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: FHI 360 (Other); Ministry of Health, Jamaica (Other); The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-6163
Record Dates: First submitted 2012-09-10; First posted 2012-09-13 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2013-04

CONDITIONS: Women Wanting Contraceptive Implant for Pregnancy Prevention
Keywords: Prostate-specific antigen; Contraceptive implant; Biological marker; Condoms; Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate implant (Experimental): Sino-implant (II) inserted at enrollment visit
  Interventions: Device: Sino-implant (II)
- Delayed implant (Active Comparator): Sino-implant (II) inserted at 3-month follow-up visit
  Interventions: Device: Sino-implant (II)

INTERVENTIONS:
Device: Sino-implant (II) — Sino-implant (II) (Shanghai Dahua Pharmaceutical Co, Ltd.; Shanghai, China), a contraceptive implant with two rods each of which contain 75 mg of levonorgestrel.
  Other Names: Zarin; TRUST; Femplant

SUMMARY:
This unblinded, randomized controlled trial (RCT) among women to determine:

1)if unprotected sex as measured prostate-specific antigen (PSA) will be more among women who receive a contraceptive implant immediately at baseline during three months of follow up compared to women who receive the implant at the three month follow-up visit.

DETAILED DESCRIPTION:
This unblinded, randomized controlled trial (RCT) will assess whether the use of a contraceptive implant leads to more sex unprotected by a condom, as measured by the detection of a biological marker of exposure to semen in vaginal fluid, among women in Kingston, Jamaica.

Eligible women will be non-pregnant, not known to be HIV-positive, 18-44 years of age, not already using a long-acting method of contraception, without contraindications to implant use, and willing to use the Sino-implant (II). Eligible women will be recruited from the Comprehensive Health Centre Center of Excellence (CHC) in Kingston, Jamaica and from the community. Women who give written consent for study participation will be enrolled in the study and randomized to one of the two study groups: 1) "immediate implant" insertion or 2) "delayed implant" insertion (i.e., when their study participation ends after three months of follow up). All participants will receive safer sex counseling, will be supplied with condoms, and will be administered a baseline questionnaire on demographics, reproductive history and contraceptive and sexual practices. A study clinician will perform a pelvic examination during which a double-headed vaginal swab will be collected to be tested for prostate-specific antigen (PSA), which is a semen biomarker. Participants will be asked to return for follow-up visits scheduled at 1 and 3 months after enrollment, at which times they will have another double-headed vaginal swab collected during a pelvic examination for testing for PSA and will be administered follow-up questionnaires. Participants in the "delayed implant" group will have the Sino-implant (II) inserted at the 3-month visit if they still want the device.

Primary objective: To determine whether the frequency of PSA detection during three months of follow up is higher in the immediate implant group than in the delayed implant group.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to be randomized to receive the implant at the enrollment visit or in three months;
* Be 18-44 years of age;
* Not known to be HIV-positive;
* Have a negative pregnancy test at baseline;
* Not currently using an intrauterine device or system, a contraceptive implant, or injectable contraception;
* Not planning to start use an intrauterine contraceptive device or system or injectable contraception in the next three months;
* Not have had surgical sterilization or plan to have it in the next three months;
* Not have medical contraindication to implant use, including lactation within first 6 weeks postpartum, acute deep venous thrombosis or pulmonary embolism, lupus, migraine with aura, unexplained vaginal bleeding, current or history of breast cancer,severe cirrhosis, liver tumors, history of stroke, and current or history of ischaemic heart disease;
* Be willing to return to the clinic for two follow-up visits over the next three months; and
* Be otherwise a good candidate for study participation based on investigator assessment

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 414 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) | 3 months
  Number of women with recent exposure to semen as measured by the detection of prostate-specific antigen (PSA) in vaginal swabs

SECONDARY OUTCOMES:
Self-reported exposure to semen | 3 months
  Number of women reporting recent exposure to semen
Side effects | 3 months
  Number of women with side effects, including changes in menstrual bleeding patterns, and mean change in body weight
Product discontinuation | 3 months
  Number of women in the immediate implant arm who discontinue implant use during the study
Acceptability | 3 months
  Number of women in the immediate implant arm who perceive the implant as acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Carole Rattray, DM, Study Chair — University of West Indies; Elizabeth Costenbader, PhD, Principal Investigator — FHI 360; Athena Kourtis, MD, PhD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Epidemiology Research Training Unit, Kingston, Kingston, Jamaica

REFERENCES:
- [Derived] Zia Y, Wiener J, Snead MC, Papp J, Phillips C, Flowers L, Medley-Singh N, Costenbader EC, Hylton-Kong T, Kourtis AP. Assessing prevalence of missed laboratory-confirmed sexually transmitted infections among women in Kingston, Jamaica: results from a secondary analysis of the Sino-Implant clinical trial. BMJ Open. 2018 Apr 13;8(4):e019913. doi: 10.1136/bmjopen-2017-019913. PMID 29654017
- [Derived] Snead MC, Wiener J, Ewumi S, Phillips C, Flowers L, Hylton-Kong T, Medley-Singh N, Legardy-Williams J, Costenbader E, Papp J, Warner L, Black C, Kourtis AP. Prevalence and risk factors associated with STIs among women initiating contraceptive implants in Kingston, Jamaica. Sex Transm Infect. 2017 Nov;93(7):503-507. doi: 10.1136/sextrans-2016-052963. Epub 2017 May 5. PMID 28476913
- [Derived] Rattray C, Wiener J, Legardy-Williams J, Costenbader E, Pazol K, Medley-Singh N, Snead MC, Steiner MJ, Jamieson DJ, Warner L, Gallo MF, Hylton-Kong T, Kourtis AP. Effects of initiating a contraceptive implant on subsequent condom use: A randomized controlled trial. Contraception. 2015 Dec;92(6):560-6. doi: 10.1016/j.contraception.2015.06.009. Epub 2015 Jun 14. PMID 26079469